CLINICAL TRIAL: NCT03051269
Title: Calcium Electroporation for Head and Neck Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Irene Wessel, Consultant, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC1511
Record Dates: First submitted 2017-01-17; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Head Neck Cancer
Keywords: Electroporation; Calcium; Head and Neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Calcium Chloride; Calcium; Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- calcium chloride (Experimental): Only one arm. All 6 enrolled patients are treated with calcium electroporation.
  Interventions: Drug: Calcium chloride; Device: Electroporation

INTERVENTIONS:
Drug: Calcium chloride — Tumour site is injected with a solution of 9 mg/ml calcium chloride and afterwards the tumour site is given electroporation to facilitate calcium to enter the cell cytosol.
  Other Names: Calcium
Device: Electroporation — Performed by single use electrodes attaches to a device called "Cliniporator" provided from IGEA, ITALY.

SUMMARY:
In a phase I protocol to primarily investigate the safety of using calcium combined with electroporation on recurrent head and neck cancers. Secondly, to evaluate tumour response on PET/MRI (positron emission tomography/magnetic resonance imaging), clinical evaluation, biopsies. Thirdly, to evaluate the effect of calcium electroporation compared to electrochemotherapy as well as the patients life-of-quality through questionnaires, EORTC QLQ C-30 and H&N35 (european organisation for research and treatment of cancer).

DETAILED DESCRIPTION:
Calcium electroporation. Electroporation is a technique that facilitates the transport of molecules across the cell membrane by using electric pulses. The electric field applied to the cell membrane creates a temporary destabilization. As the electric capacity of the membrane is exceeded, cracks are formed in the membrane and the molecules are free to diffuse into the cytosol of the cell. The process is reversible and the cell membrane is stabilized in a matter of minutes. While the cell membrane is permeable there is an increased influx of Ca2+ into the cell. Calcium influx may be further improved by combining calcium together with electroporation; this is called calcium electroporation.

In vivo studies have shown that when enhancing the extracellular calcium concentration before applying electroporation, a larger Ca2+ influx occurs. The large Ca2+ influx can lead to a reduction in ATP (adenosine triphosphate) levels and cell death. A fall in ATP levels is seen for two reasons: First, an increase in intracellular Ca2+ leads to a higher activity of the Ca2+-ATPase and Na+/K+-ATPase. Secondly, the high concentration of Ca2+ leads to loss of the electrochemical gradient in the mitochondrial membrane, which causes mitochondrial collapse. Upon collapse of the mitochondria, the cell can no longer produce ATP. Overall, the increased consumption and decreased production of ATP leads to lover ATP levels. Combined with other cellular processes such as activation of lipases and proteases, the cell will eventually die.

Trials objectives.

1. Primary outcome. Evaluating the safety measures of using calcium electroporation on mucosal head and neck cancer. This is done by continuously evaluating pain by VAS-score (visual analogue scale) and side effects by Common Terminology Criteria for Adverse Events (CTCAE) registration into Adverse Events (AE) and Serious Adverse Events (SAE). The safety of using calcium intratumourally is also evaluated by measurement of Ca2+ in blood samples after treatment.
2. Secondary outcome. Evaluation of response by imaging: PET-MRI, Clinical photography, Biopsies from tumour site The subjects subjective evaluation of the treatment and post treatment period is evaluated through Quality of life questionnaires, EORTC QLQ-C30 and H&N35: two different questionnaires both validated for head and neck cancer patients.
3. Tertiary outcome. The response to treatment will be compared to the results from our current trial, where we use electrochemotherapy on mucosal head and neck tumours. The comparison will be between imaging response, VAS score and results from questionnaires (EORTC QLQ-C30 and H&N35).

Trial design. This is a phase I, interventional, clinical trial for the safety of calcium electroporation on mucosal head and neck tumours. Subjects will have relapsed or primary head and neck cancer. Treatment is intended as palliative and not curative. All subjects will be offered standard treatment with surgery and radiotherapy before enrolment to the trial, if possible. There is no scheduled control group, meaning that all eligible patients will be offered treatment.

Electroporation and anaesthesia. The treatment is performed under general anaesthesia because the localization of head and neck tumours complicates treatment under local anaesthetic. After the patient is anaesthetized, the tumour area will be injected with calcium. After administration of calcium electrodes are inserted into the tumour and electrical pulses are generated and documented using a Cliniporator (IGEA, Capri, Italy). Overall operating time/anaesthesia time will be 1-2 hours and expected hospital stay of 3 days. Treatment is intended as a once-only treatment but measurable response on evaluation scans combined with continued cancer activity in the treated area can result in another treatment session.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age > 18 years.
2. Verified cancer in the head and neck region of any histology.
3. At least one tumour lesion should be accessible for electroporation.
4. Performance status WHO <= 2.
5. Progressive and/or metastatic disease.
6. Expected survival of > 3 months.
7. A treatment-free interval of more than 4 weeks since chemotherapy or radiation therapy of the treatment area.
8. The subject should have been offered the current standard treatment. If there is no further standard treatment to offer or if the subject does not want to receive the treatments offered, the subject may be included in the trial.
9. The subject should be able to understand the information for participants and be willing and able to comply with hospitalization and the agreed follow-up visits and tests.
10. Platelets ≥ 50 billion/L, INR(international normalized ratio)> 1.5. Medical correction is allowed, e.g. correction of a high INR using vitamin K.
11. Sexually active men and women who can become pregnant must use adequate contraception during this trial (pill, spiral, injection of prolonged progestin, subdermal implantation, hormone-containing vaginal devices, transdermal patches).
12. Signed informed consent.

    -

Exclusion Criteria:

Patients should be excluded if they meet just one of the criteria stated below:

1. Symptomatic progression of the subject's cancer disease that requires another intervention.
2. Allergy to constituents of the planned anesthesia.
3. Coagulation disorder that cannot be corrected.
4. Chronic renal dysfunction with creatinine> 200 mmol/L will trigger a Cr-51-EDTA (Ethylenediaminetetraacetic acid) clearance.
5. Pregnancy or lactation.
6. If participating in other clinical trials involving experimental drugs or involved in a trial within 4 weeks prior to study drug administration.
7. Other disorders investigator finds incompatible with participation in the trial.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change in Treatment-Emergent Adverse Events [Safety and Tolerability] | CTCAE are evaluated at several timepoints: 1) Baseline (before treatment). 2) 30 minutes and 6 hours after treatment. 3) Once at day 1, 2 and 3 after treatment. 4) 1 week after treatment. 5) 2 weeks after treatment. 6) 1 and 2 months after treatment.
  Evaluated by change in CTCAE (common terminology criteria for adverse events) at different timepoints.
Change in Treatment-Emergent Adverse Events [Safety and Tolerability] | Blood samples evaluating calcium levels are taken at 1) Baseline. 2) 30 min after treatment. 3) 6 hours after treatment. 4) At day 1, 2, and 3 after treatment.
  Evaluated by change in calcium levels in blood samples at different time points.

SECONDARY OUTCOMES:
Tumour response | PET/MRI are performed at baseline and evaluated again at 1 and 2 months after treatment.
  By PET/MRI imaging
Tumour response | Clinical evaluation is performed daily in the first 3 days post-treatment, again at week 1 and 2, and 1 and 2 months post-treatment.
  By clinical evaluation.
Tumour response | Biopsies are performed at baseline and again at 1 and 2 months after treatment.
  By biopsies.
Comparing calcium electroporation to electrochemotherapy | 1 year
  The tumor response on MRI from calcium electroporation is compared to the tumor response on MRI from a previous study on a similar patient group treated with electrochemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Wessel, Principal Investigator — Rigshospitalet, Dept. of Head and Neck Surgery, Copenhagen, Denmark
Locations (1):
- Department of Otorhinolaryngology, Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frandsen SK, Gibot L, Madi M, Gehl J, Rols MP. Calcium Electroporation: Evidence for Differential Effects in Normal and Malignant Cell Lines, Evaluated in a 3D Spheroid Model. PLoS One. 2015 Dec 3;10(12):e0144028. doi: 10.1371/journal.pone.0144028. eCollection 2015. PMID 26633834
- [Background] Hansen EL, Sozer EB, Romeo S, Frandsen SK, Vernier PT, Gehl J. Dose-dependent ATP depletion and cancer cell death following calcium electroporation, relative effect of calcium concentration and electric field strength. PLoS One. 2015 Apr 8;10(4):e0122973. doi: 10.1371/journal.pone.0122973. eCollection 2015. PMID 25853661
- [Background] Frandsen SK, Gissel H, Hojman P, Tramm T, Eriksen J, Gehl J. Direct therapeutic applications of calcium electroporation to effectively induce tumor necrosis. Cancer Res. 2012 Mar 15;72(6):1336-41. doi: 10.1158/0008-5472.CAN-11-3782. Epub 2012 Jan 26. PMID 22282658
- [Background] Plaschke CC, Gothelf A, Gehl J, Wessel I. Electrochemotherapy of mucosal head and neck tumors: a systematic review. Acta Oncol. 2016 Nov;55(11):1266-1272. doi: 10.1080/0284186X.2016.1207803. Epub 2016 Oct 5. PMID 27705053